CLINICAL TRIAL: NCT02777294
Title: Evaluation of Web-Based CBT for Rape Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Boston University (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Heather Littleton, Associate Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH085118-01A2 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online intervention (Experimental): Therapist-facilitated, cognitive behavioral therapy
  Interventions: Behavioral: Online intervention
- Psycho-educational website (Active Comparator): Self-help, psycho-educational website
  Interventions: Behavioral: Psycho-educational website

INTERVENTIONS:
Behavioral: Online intervention — Therapist-facilitated, multimedia, cognitive-behavioral online intervention targeting rape-related PTSD
  Arms: Online intervention
Behavioral: Psycho-educational website — Psycho-educational self-help website about rape-related PTSD
  Arms: Psycho-educational website

SUMMARY:
Rape is unfortunately a common experience among women, affecting between 13 and 20%. In addition, up to 50% of all rape victims experience significant and persistent psychological distress. While cognitive-behavioral interventions have been found to be successful at alleviating distress among victims; the majority do not seek out these services, often because of feelings of stigma and self-blame. One potential method for circumventing these barriers is through online administered treatment. Thus, the current project is designed to conduct an initial evaluation of a 12 to 16-week, therapist-facilitated, multi-media, cognitive-behavioral, online intervention tailored specifically for rape victims. The effectiveness of this program at ameliorating distress among college women who have experienced rape and have current posttraumatic stress disorder (PTSD) was evaluated. Reductions in psychological distress was the primary outcome and was assessed at post-intervention and at three and six month follow-up periods. The effectiveness of the intervention was compared to a psycho-educational website.

ELIGIBILITY:
Inclusion Criteria:

* Current rape-related PTSD
* Regular access to a computer
* English language literacy
* Experience of completed rape at age 14 years or older

Exclusion Criteria:

* No current PTSD
* Current psychotherapy
* Lack of stability on psychotropic medication (< 3 months)
* Lack of literacy in English
* Current substance dependence
* Current elevated suicidality
* Severe acute distress
* No experience of completed rape after age 14

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms (PTSD Symptom Scale Interview) | Change in PTSD symptoms from baseline to 3 months post intervention

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783